CLINICAL TRIAL: NCT06669442
Title: The Effectiveness of Guided Imagery, a Mindfulness Technique, on PCL-5 Scores in Adult Women With Post-Traumatic Stress Disorder
Brief Title: The Effectiveness of Guided Imagery on PCL-5 Scores in Adult Women With Post-Traumatic Stress Disorder
Acronym: PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Kellie-Ann Kerr, Principal Investigator, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-471
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-04

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: Guided Imagery; Mindfulness; Post Traumatic Stress Disorder; Adult Women; Women; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guided Imagery Mindfulness (Experimental): Mindfulness-based interventions (MBIs), such as guided imagery, emerge as promising alternatives for managing PTSD. Mindfulness necessitates participant training to maintain present awareness amidst wandering thoughts, fostering an attitude of non-judgmental acceptance towards thoughts and emotions. Mindfulness encourages, being present in the moment and supports emotional control.
  Interventions: Behavioral: Guided Imagery

INTERVENTIONS:
Behavioral: Guided Imagery — Guided imagery is a mindfulness based therapeutic technique that involves utilizing positive imagery allowing one to cultivate awareness of their mental state and shift their attention from ruminative thought patterns to the present moment. Evidence-based research shows that benefits of Guided imagery include relaxation, stress reduction, anxiety reduction, immune system enhancement, and overall well-being.
  Other Names: Guided Meditation; Visualization; Imagery; Mental Imagery; Mental Rehearsal

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) affects a significant portion of the population, with about 13 million Americans diagnosed in 2020. Women are twice as likely to have PTSD than men. PTSD will affect 8%, or 8 out of every 100 women, at some stage in their lives. This study will check the effects of guided imagery mindfulness on PCL-5 scores in adult women with PTSD. Participants in this study will complete a PCL-5 pre-test and post-test to check PTSD symptoms before and after 6-weeks of mindfulness sessions. Each participant will engage in 15-minute sessions of guided imagery mindfulness once a week for 6 weeks. Before and after PCL-5 scores will show the effect of guided imagery mindfulness on PTSD symptom severity.

DETAILED DESCRIPTION:
Background: Post-Traumatic Stress Disorder (PTSD) affects a significant portion of the population, with approximately 13 million Americans diagnosed in 2020. Women are twice as likely to have PTSD than men. PTSD will affect 8%, or 8 out of every 100 women, at some stage in their lives.

Purpose: This project aims to investigate the effectiveness of guided imagery, a mindfulness technique, on PCL-5 scores in adult women with PTSD.

Theoretical Framework: The Cognitive model of PTSD was developed to explain why some people do not recover after trauma and to identify maintaining factors that can be modified in treatment. This model suggests negative appraisals, disjointed trauma memories, and unhelpful coping strategies maintain PTSD.

Methods: Participants in this qualitative study will complete pre- and post-intervention PCL--5 questionnaires, a validated 20-item structured interview designed to assess PTSD symptoms. They will also engage in 15-minute sessions of guided imagery mindfulness interventions. Post-intervention, participants will complete a second PCL-5 questionnaire to evaluate any changes in symptom severity.

Results: Analysis of PCL-5 scores will provide insight into the effect of guided imagery mindfulness interventions on PTSD symptom severity.

Conclusions: Mindfulness has the potential to serve as a viable alternative or supplemental intervention for women diagnosed with PTSD. Through exploring the potential benefits of mindfulness-based interventions in managing PTSD symptoms, this study seeks to aid in the advancement of more effective treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Females
* PTSD diagnosis (ICD 10: F43.1)
* 18 to 99 years old
* Not pregnant
* No suicidal ideations
* No homicidal ideations
* No audio-visual hallucinations
* A mobile device, smart phone, laptop
* Resident at the Residential Treatment Facility

Exclusion Criteria:

* Males
* Under 18 years old
* Above 99 years old
* Pregnant women
* Active suicidal ideation
* Active homicidal ideation
* Do not have mobile device
* Active audio-visual hallucinations

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 15 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline PTSD Symptom Severity Using PTSD Checklist for DSM-5 (PCL-5) Scores at 6 weeks | 6 weeks
  PCL-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms.
  Participants rate how bothered they have been by each of 20 items in the past month on a 5- point Likert scale ranging from 0-4.
  Items are summed to provide a total severity score (range = 0-80). 0 = Not at all 1 = A little bit 2 = Moderately 3 = Quite a bit 4 = Extremely
  Range: 0 (best outcome) to 80 (worst outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Jessie Trice Community Health Systems, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect the privacy and confidentiality of the participants. Sharing participant data may pose risks of identifying individuals in studies, with limited sample sizes or unique demographic profiles.

REFERENCES:
- [Background] Waldron EM, Burnett-Zeigler I. The impact of participation in a mindfulness-based intervention on posttraumatic stress symptomatology among Black women: A pilot study. Psychol Trauma. 2022 Jan;14(1):29-37. doi: 10.1037/tra0001107. Epub 2021 Aug 26. PMID 34435817
- [Background] Saban KL, Collins EG, Mathews HL, Bryant FB, Tell D, Gonzalez B, Bhoopalam S, Chroniak CP, Janusek LW. Impact of a Mindfulness-Based Stress Reduction Program on Psychological Well-Being, Cortisol, and Inflammation in Women Veterans. J Gen Intern Med. 2022 Sep;37(Suppl 3):751-761. doi: 10.1007/s11606-022-07584-4. Epub 2022 Aug 30. PMID 36042095
- [Background] Roberts NP, Kitchiner NJ, Lewis CE, Downes AJ, Bisson JI. Psychometric properties of the PTSD Checklist for DSM-5 in a sample of trauma exposed mental health service users. Eur J Psychotraumatol. 2021 Jan 26;12(1):1863578. doi: 10.1080/20008198.2020.1863578. eCollection 2021. PMID 34992744
- [Background] McNicholas C, Lennox L, Woodcock T, Bell D, Reed JE. Evolving quality improvement support strategies to improve Plan-Do-Study-Act cycle fidelity: a retrospective mixed-methods study. BMJ Qual Saf. 2019 May;28(5):356-365. doi: 10.1136/bmjqs-2017-007605. Epub 2019 Mar 18. PMID 30886118
- [Background] Kozlov E, Bantum E, Pagano I, Walser R, Ramsey K, Taylor K, Jaworski B, Owen J. The Reach, Use, and Impact of a Free mHealth Mindfulness App in the General Population: Mobile Data Analysis. JMIR Ment Health. 2020 Nov 27;7(11):e23377. doi: 10.2196/23377. PMID 33245289
- [Background] Krau SD. The Multiple Uses of Guided Imagery. Nurs Clin North Am. 2020 Dec;55(4):467-474. doi: 10.1016/j.cnur.2020.06.013. Epub 2020 Oct 14. PMID 33131625
- [Background] Kachadourian LK, Harpaz-Rotem I, Tsai J, Southwick S, Pietrzak RH. Mindfulness as a mediator between trauma exposure and mental health outcomes: Results from the National Health and Resilience in Veterans Study. Psychol Trauma. 2021 Feb;13(2):223-230. doi: 10.1037/tra0000995. Epub 2021 Jan 21. PMID 33475404
- [Background] Haider T, Dai CL, Sharma M. Efficacy of Meditation-Based Interventions on Post-Traumatic Stress Disorder (PTSD) Among Veterans: A Narrative Review. Adv Mind Body Med. 2021 Winter;35(1):16-24. PMID 33513582
- [Background] Gibson J. Trauma, early life stress, and mindfulness in adulthood. BMC Psychol. 2024 Feb 14;12(1):71. doi: 10.1186/s40359-024-01563-6. PMID 38355582
- [Background] Ehlers A, Grey N, Wild J, Stott R, Liness S, Deale A, Handley R, Albert I, Cullen D, Hackmann A, Manley J, McManus F, Brady F, Salkovskis P, Clark DM. Implementation of cognitive therapy for PTSD in routine clinical care: effectiveness and moderators of outcome in a consecutive sample. Behav Res Ther. 2013 Nov;51(11):742-52. doi: 10.1016/j.brat.2013.08.006. Epub 2013 Sep 10. PMID 24076408
- [Background] Beierl ET, Bollinghaus I, Clark DM, Glucksman E, Ehlers A. Cognitive paths from trauma to posttraumatic stress disorder: a prospective study of Ehlers and Clark's model in survivors of assaults or road traffic collisions. Psychol Med. 2020 Oct;50(13):2172-2181. doi: 10.1017/S0033291719002253. Epub 2019 Sep 11. PMID 31507261
- See also: Mindfulness Coach App — https://www.ptsd.va.gov/appvid/mobile/mindfulcoach_app.asp
- See also: PTSD Checklist for DSM-5 (PCL-5) — https://www.ptsd.va.gov/professional/assessment/documents/PCL5_Standard_form.PDF